CLINICAL TRIAL: NCT07009470
Title: A Multicenter, Prospective Study of Perioperative Finotonlimab Combined With Bevacizumab in Resectable Hepatocellular Carcinoma Patients With High-Risk Factors for Recurrence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhiyong Huang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-SCT-TJ01
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-02

CONDITIONS: HCC
Keywords: adjuvant regimen; TACE combined with targeted-immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined with targeted-immunotherapy (Experimental)
  Interventions: Drug: Finotonlimab (an anti-PD-1 monoclonal antibody) and Anbeizhu (a bevacizumab biosimilar); Procedure: TACE

INTERVENTIONS:
Drug: Finotonlimab (an anti-PD-1 monoclonal antibody) and Anbeizhu (a bevacizumab biosimilar) — First, perform a single session of TACE. Followed by three cycles of neoadjuvant therapy with Finotonlimab combined with bevacizumab. Proceed with curative resection. Finally, initiate postoperative adjuvant targeted-immunotherapy . Finotonlimab: intravenously every three weeks ,200mg. bevacizumab：intravenously every three weeks , with a dosage based on body weight: 15 mg (≤60 kg) .
Procedure: TACE — Initial Perform a single session of TACE procedure.TACE treatment is strictly in accordance with the Chinese guidelines for clinical practice of transcatheter arterial chemoembolization (TACE) for hepatocellular carcinoma (2023 Edition).

SUMMARY:
For patients with early- to mid-stage hepatocellular carcinoma (HCC), the five-year postoperative recurrence and metastasis rate remains as high as 70%, significantly impacting patient prognosis.Therefore, perioperative therapy may be considered for HCC patients with these high-risk features .

ELIGIBILITY:
Inclusion Criteria:

1. - Informed Consent Voluntarily signed informed consent after full understanding of the study, with commitment to comply with all protocol requirements and assessment schedules.
2. Age 18-75 years inclusive.
3. Diagnosis Histologically/cytologically confirmed hepatocellular carcinoma (HCC) OR clinically diagnosed HCC per 2024 Chinese Guidelines for Primary Liver Cancer.
4. Tumor Status

   Meets ONE of the following:

   Multifocal tumors (2-4 lesions)

   Single lesion >5 cm in longest diameter

   Stage IIIa HCC with Vp1/Vp2/Vp3 portal vein tumor thrombus
5. Resectability Technically amenable to curative resection per surgeon assessment.
6. Liver Function Child-Pugh class A.
7. Performance Status ECOG PS 0-1.
8. Prior Therapy No previous systemic treatment for HCC.
9. Measurable Disease

   ≥1 radiologically measurable lesion per mRECIST.
10. Organ Function (1) Hematological:

    ANC ≥1.5×10⁹/L

    Hemoglobin ≥90 g/L

    Platelets ≥50×10⁹/L (2) Hepatic:

    Total bilirubin ≤1.5×ULN

    AST/ALT ≤2.5×ULN

    Albumin ≥28 g/L (3) Coagulation:

    INR ≤2.3 OR PT prolongation ≤3 sec vs control (4) Renal:

    eGFR >90 mL/min/1.73m² (CKD-EPI)
11. Contraception

Women of childbearing potential: Negative serum pregnancy test within 7 days prior to enrollment.

All subjects: Use highly effective contraception during treatment and for 180 days post-last dose.

Exclusion Criteria:

1. Pregnancy/Lactation Women who are pregnant or breastfeeding.
2. Concurrent Malignancy

   History of other malignancies within 5 years except:
3. Curatively treated basal cell carcinoma

   Cervical carcinoma in situ

   Papillary thyroid carcinoma
4. Drug Hypersensitivity Known allergy to finolizumab, bevacizumab, or their excipients.

   Bleeding Risk History of upper GI bleeding OR active hemorrhagic disorders.
5. Uncontrolled Cardiac Disease

   Clinically significant cardiac conditions including:

   NYHA Class II+ heart failure

   Unstable angina

   Myocardial infarction within 1 year

   Clinically significant arrhythmias requiring intervention
6. Autoimmune Disorders Active autoimmune diseases or history of autoimmune disorders.
7. Immunodeficiency

   Immunodeficiency conditions including:

   HIV positive status

   Primary/secondary immunodeficiency

   History of organ/bone marrow transplantation
8. Psychiatric Conditions Severe psychiatric disorders OR substance abuse involving psychotropic drugs.
9. Uncontrolled Comorbidities Severe uncontrolled recurrent infections OR other significant uncontrolled comorbidities.
10. Investigator Discretion Any condition deemed ineligible by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2028-04-28 (Estimated); Study Completion 2028-10-28 (Estimated)

PRIMARY OUTCOMES:
2-year DFS rate and 2-year OS rate | 2years
  2-year DFS rate refers to the proportion of patients remaining free of disease recurrence or death for over 2 years, measured from the date of surgery.
  2-year OS rate refers to the proportion of subjects surviving in the trial cohort at the 2-year follow-up mark, calculated from the initiation of neoadjuvant therapy.

SECONDARY OUTCOMES:
MPR | 9 weeks
  Defined as the presence of ≥70% tumor necrosis in the tumor bed and regional lymph nodes of resected specimens following curative resection.
pCR | 9 weeks
  Defined as the absence of viable tumor cells in both the primary tumor site and regional lymph nodes of resected specimens after curative surgery.
R0 rate | 9 weeks
  The tumor was completely removed with negative margins, meaning no residual tumor
EFS | 2 years
  Event Free Survival
safety | 2 years
  Safety profiles during neoadjuvant therapy and postoperative period were systematically assessed per CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Huang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No